CLINICAL TRIAL: NCT03350178
Title: Evaluation of Heterologous Fecal microbiotA Transfer in ICU Patients: a FeasibilitY and SafetY StudY
Acronym: HAPY3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment shortened
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MPICU01
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Intensive Care Units; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated patients (Experimental): Treated wit FMT
  Interventions: Drug: fecal microbiota transfer

INTERVENTIONS:
Drug: fecal microbiota transfer — transfer of fecal microbiota from healthy donor to the patients

SUMMARY:
ICU patient's complications are notably due to multiple infections with high risks of sepsis. Those infections would be worsened by any antibiotic resistance mechanism. Thus, reducing MDR portage in health care unit is a global strategy that will benefit for the patients and the health system organization. Fecal Microbiota transfer and restoration is a promising strategy to achieve this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients hospitalized in ICU
* Patients under mechanical ventilation
* Patients with an expected length of stay of at least 4 days after inclusion
* Patients identified with an MDRB digestive carriage, determined by a positive rectal swab previously performed during ICU stay, according to usual screening
* Expected antibiotic (ATB) duration < 10 days
* Informed written consent from the patient
* In unconscious patients who are not able to give consent for inclusion in the study, relatives (next-of-kin) give assent on every patient's behalf, and patients will be later given the opportunity to withdraw from the study

Exclusion Criteria:

* Patients with a high risk of death within 5 days according to investigator's opinion, or subjected to therapeutic limitation decisions
* Antibiotherapy of more than 4 consecutive days at inclusion
* Confirmed or suspected intestinal ischemia
* Confirmed or suspected toxic megacolon or gastrointestinal perforation
* Any gastro-intestinal bleeding in the past 3 months
* Any history of abdominal surgery in the past 3 months
* Any history of chronic digestive disease or gastro-intestinal resection
* Any counter indication for Trendelenburg position
* Neutropenia (neutrophil counts < 500 cells/µL)
* Ongoing immunosuppressive therapy (chemotherapy, any immunosuppressive agents, excluding corticosteroids < 0,5 mg/kg/d of equivalent prednisolone)
* Enrollment in another trial that may interfere with this study
* Known allergy or intolerance to trehalose or maltodextrin and latex
* Pregnancy or breastfeeding
* Patients with EBV- serology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of FMT-related treatment emergent (serious) adverse events | through study completion, an average of 2 weeks
  Occurrence of FMT-related treatment emergent (serious) adverse events

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 2 weeks
  FMT procedure will be considered as good if it has been accepted without any particular reluctance
Occurrence of FMT-related treatment emergent (serious) adverse events as per investigator's opinion | through study completion, an average of 2 weeks
  occurrence of FMT-related treatment emergent (serious) adverse events
Evaluation of FMT impact on Multi Drug Resistant Bacteria carriage | through study completion, an average of 2 weeks
  Based on bacterial culture, description of MDRB carriage. Resistance acquisition or eradication will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Rouze, Principal Investigator — CHRU LILLE
Locations (2):
- France (2):
  - Salengro hospital, Lille
  - Bichat Hospital, Paris

IPD SHARING:
Plan to Share IPD: No